CLINICAL TRIAL: NCT01688635
Title: Comparative Pharmacokinetics and Pharmacodynamics of LY2963016 and US-Approved Lantus® After Single-Dose Subcutaneous Administration to Healthy Subjects
Brief Title: A Study to Compare LY2963016 and US-approved Lantus® After Single Dose Administration to Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14973; I4L-MC-ABEO (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-09-17; First posted 2012-09-20 (Estimated); Results first posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Volunteers
MeSH Terms: interventions — LY2963016 insulin glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- LY2963016 (Experimental): Single 0.5 units per kilogram (U/kg) dose of LY2963016 administered subcutaneously, twice during the study
  Interventions: Drug: LY2963016
- US-approved Lantus (Experimental): Single 0.5 U/kg dose of US-approved Lantus administered subcutaneously, twice during the study
  Interventions: Drug: US Approved Lantus

INTERVENTIONS:
Drug: LY2963016 — Administered subcutaneously
  Arms: LY2963016
Drug: US Approved Lantus — Administered subcutaneously
  Arms: US-approved Lantus

SUMMARY:
The purpose of this study is to compare the pharmacokinetics and pharmacodynamics of LY2963016 and US-approved Lantus®. The study involves four single injections; two doses of LY2963016 and two doses of US-approved Lantus®. The study will have 4 periods. In each period, a single injection will be administered before undergoing a euglycemic clamp that lasts for 24 hours. There will be at least a 7 day washout between each period. Side effects will be documented. Study participation is expected to last up to 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females
* Have body mass index between 18.5 and 29.9 kilograms per meter square (kg/m^2)
* Are nonsmokers and have not smoked for at least 2 months prior to entering the study
* Have normal blood pressure and pulse rates at screening
* Have electrocardiograms (ECGs) at screening considered as within normal limits
* Have clinical laboratory test results within normal reference ranges

Exclusion Criteria:

* Are currently enrolled in or discontinued within the last 30 days from a clinical study involving an investigational drug or device or are concurrently enrolled in any other type of medical research
* Have known allergies to insulin, its excipients, or related drugs or have history of relevant allergic reactions of any origin
* Have significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders
* Show evidence of significant active neuropsychiatric disease, including taking prescription medication for such diseases
* Show evidence of current use of known drugs of abuse or a history of use within the past year
* Have a history of first-degree relatives known to have diabetes mellitus
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies at screening
* Have positive hepatitis B surface antigen at screening
* Intend to use over-the-counter or prescription medication within 7 or 14 days, respectively, prior to dosing (apart from vitamin/mineral supplements, occasional paracetamol, thyroid replacement medication, or birth control methods)
* Have donated or had a blood loss of 450 milliliters (mL) within 3 months prior to study enrollment
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females) or are unwilling to stop alcohol consumption from 24 hours prior to each dosing until discharged from the clinical research unit (CRU)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2012-09; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study comprised 2 sequences with 4 treatment periods. Participants were randomly assigned to 1 of the 2 sequences.
Groups:
- LY/Lantus/LY/Lantus: A single 0.5-units/kilogram (U/kg) dose of LY2963016 (LY) administered subcutaneously during Periods 1 and 3.
  A single 0.5-U/kg dose of US-approved Lantus (Lantus) administered subcutaneously during Periods 2 and 4.
  There was at least a 7-day washout between treatment periods.
- Lantus/LY/Lantus/LY: A single 0.5-U/kg dose of US-approved Lantus administered subcutaneously during Periods 1 and 3.
  A single 0.5-U/kg dose of LY2963016 administered subcutaneously during Periods 2 and 4.
  There was at least a 7-day washout between treatment periods.
Period: Period 1
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 45 | 46
Received at Least 1 Dose of Study Drug | 45 | 46
Completed | 45 | 46
Not Completed | 0 | 0
Period: Washout 1
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 45 | 46
Completed | 44 | 44
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 0 | 1
Period: Period 2
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 44 | 44
Completed | 44 | 44
Not Completed | 0 | 0
Period: Washout 2
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 44 | 44
Completed | 41 | 42
Not Completed | 3 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Sponsor Decision | 1 | 2
Period: Period 3
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 41 | 42
Completed | 41 | 42
Not Completed | 0 | 0
Period: Washout 3
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 41 | 42
Completed | 40 | 42
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 4
Arm/Group | LY/Lantus/LY/Lantus | Lantus/LY/Lantus/LY
Started | 40 | 42
Completed | 40 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- LY2963016 and US-approved Lantus: Single 0.5-units per kilogram (U/kg) dose of LY2963016 administered subcutaneously twice during the study; Single 0.5-U/kg dose of US-approved Lantus administered subcutaneously twice during the study. There was at least a 7-day washout between treatment periods.
Arm/Group | LY2963016 and US-approved Lantus
Number analyzed (Participants) | 91
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.7 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 85
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 90
  White | 1
Region of Enrollment [Number; unit: participants]
  Singapore | 91

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under the Concentration Time Curve (AUC) of LY2963016 and US-Approved Lantus
Description: The AUC from time 0 to 24 hours (AUC0-24) of LY2963016 and US-Approved Lantus was measured.
Time Frame: 30 minutes predose up to 24 hours postdose in all treatment periods
Population: Full analysis set (FAS): All randomized participants who received at least 1 dose of study drug and had evaluable PK data to calculate AUC(0-24). Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles*hour/liter (pmol*h/L)
Groups:
- LY2963016: Single 0.5-units per kilogram (U/kg) dose of LY2963016 administered subcutaneously twice during the study. There was at least a 7-day washout between treatment periods.
- US-approved Lantus: Single 0.5-U/kg dose of US-approved Lantus administered subcutaneously twice during the study.
  There was at least a 7-day washout between treatment periods.
Arm/Group | LY2963016 | US-approved Lantus
Number analyzed (Participants) | 87 | 89
picomoles*hour/liter (pmol*h/L) | 1720 (42) | 1900 (35)

2. Primary Outcome: Pharmacokinetics (PK): Maximum Plasma Concentration (Cmax) of LY2963016 and US-Approved Lantus
Time Frame: 30 minutes predose up to 24 hours postdose in all treatment periods
Population: Full analysis set (FAS): All randomized participants who received at least 1 dose of study drug and had evaluable PK data to calculate Cmax. Participants were analyzed based on the treatment they received
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomoles/liter (pmol/L)
Arm/Group | LY2963016 | US-approved Lantus
Number analyzed (Participants) | 88 | 89
picomoles/liter (pmol/L) | 103 (41) | 111 (34)

3. Secondary Outcome: Maximum Glucose Infusion Rate (Rmax)
Description: Rmax is the maximum infusion rate of glucose administered intravenously needed to maintain target blood glucose level and is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of LY2963016 or US-approved Lantus by adjusting the exogenous glucose infusion rate. Data presented were adjusted by the body weight.
Time Frame: 30 minutes predose up to 24 hours postdose in all treatment periods
Population: Full analysis set (FAS): All randomized participants who received at least 1 dose of study drug and had evaluable pharmacodynamic data to calculate Rmax. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilograms/minute (mg/kg/min)
Arm/Group | LY2963016 | US-approved Lantus
Number analyzed (Participants) | 88 | 88
milligrams/kilograms/minute (mg/kg/min) | 2.12 (54) | 2.27 (58)

4. Secondary Outcome: Total Amount of Glucose Infused (Gtot) Over the Duration of Clamp Procedure
Description: Gtot was the total glucose infusion over the clamp duration and was used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations were held constant after the administration of LY2963016 or US-approved Lantus by adjusting the exogenous glucose infusion rate. Data presented were adjusted by the body weight.
Time Frame: 30 minutes predose up to 24 hours postdose in all treatment periods
Population: Full analysis set (FAS): All randomized participants who received at least 1 dose of study drug and had evaluable pharmacodynamic data to calculate Gtot. Participants were analyzed based on the treatment they received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilogram (mg/kg)
Arm/Group | LY2963016 | US-approved Lantus
Number analyzed (Participants) | 88 | 88
milligrams/kilogram (mg/kg) | 1670 (60) | 1820 (74)

ADVERSE EVENTS:
Time Frame: Randomization to study completion
Description: Study-specific clinical outcomes due to progressive disease were not considered to be serious adverse events (SAEs) unless it was deemed related to study drug by the investigator.
Groups:
- LY2963016: Single 0.5 units per kilogram (U/kg) dose of LY2963016 administered subcutaneously twice during the study.
  There was at least a 7-day washout between the treatment periods.
- US-approved Lantus: Single 0.5 U/kg dose of US-approved Lantus administered subcutaneously twice during the study.
  There was at least a 7-day washout between the treatment periods.
Arm/Group | LY2963016 | US-approved Lantus
Serious Adverse Events (participants affected / at risk) | 0/89 | 0/90
Other Adverse Events (participants affected / at risk) | 42/89 | 42/90
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2963016 (N=89) | US-approved Lantus (N=90)
Catheter site haematoma (General disorders) | 10 (11) | 9 (11)
Catheter site pain (General disorders) | 5 (5) | 6 (6)
Catheter site swelling (General disorders) | 9 (10) | 7 (7)
Infusion site pain (General disorders) | 4 (4) | 4 (5)
Infusion site swelling (General disorders) | 2 (2) | 5 (6)
Pyrexia (General disorders) | 4 (4) | 1 (1)
Procedural site reaction (Injury, poisoning and procedural complications) | 2 (2) | 4 (5)
Headache (Nervous system disorders) | 3 (3) | 8 (9)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes